CLINICAL TRIAL: NCT01404793
Title: The Use Of Solid Phase Micro Extraction For Metabolomic Profiling And Concomitant Measurements Of Rocuronium Bromide Levels In Recipients Of Orthotopic Liver Transplantations
Brief Title: SPME For Metabolomics And Concomitant Measurements Of Rocuronium Bromide Levels In Liver Transplantation
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 11-0325-BE
Record Dates: First submitted 2011-07-26; First posted 2011-07-28 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Liver Failure
Keywords: Liver Transplantation; Solid Phase Micro Extraction; Rocuronium; Metabolomics; Pharmacokinetics; Clinical Marker
MeSH Terms: conditions — Liver Failure | interventions — Rocuronium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver transplant recipient
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium — After insertion of the new liver and restoration of portal venous flow, 0.6 mg kg-1 rocuronium will be administered
  Other Names: Zemuron; Esmeron

SUMMARY:
Standard anesthetic management of liver transplantation patients includes a general anesthetic using multiple drugs, including the neuromuscular relaxant rocuronium. Pharmacokinetic modelling of this agent has been poorly described during liver transplantation, which impacts on appropriate dosing of this agent within this population where plasma concentrations can vary with fluid shifts and hepatic drug metabolism during the various phases of liver transplantation. Plasma drug and drug metabolite concentrations will be measured using the technique of solid phase micro-extraction (SPME). Measuring and correlating the levels of rocuronium and other liver metabolites with the degree of post transplantation hepatic dysfunction may serve as a simple and cost-effective marker to aid diagnosis, identify those at risk of hepatic dysfunction and potentially grade the severity

ELIGIBILITY:
Inclusion Criteria:

* First time liver transplant recipients above 18 years of age
* Elective cadaveric or living donor liver transplant patients will be recruited

Exclusion Criteria:

* All patients under 18 years of age
* Unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving liver transplants at University Health Network, Toronto General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Plasma drug and drug metabolite concentrations | 5, 30, 60, 90, 120, 180, 240, 300, 450 mins
  All liver transplant recipients in this study will receive standard level of care including general anesthesia and the use of invasive arterial and central line monitoring. On induction, patients will receive the neuromuscular relaxant cisatracurium at 0.1 mg kg-1. After insertion of the new liver and restoration of portal venous flow, 0.6 mg kg-1 rocuronium will be administered. If further muscle relaxation is required, cistaracurium will be administered. Collection of 5ml blood samples will be performed at: 5, 30, 60, 90, 120, 180, 240, 300, 450 mins post bolus administration.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Wasowicz, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada